CLINICAL TRIAL: NCT00483509
Title: NGR007: A Phase II Study of NGR-hTNF Administered in Combination With Doxorubicin Every 3 Weeks in Patients Affected by Advanced or Metastatic Small Cell Lung Carcinoma (SCLC) Previously Treated With at Least One Therapeutic Regimen
Brief Title: Study of NGR-hTNF in Combination With Doxorubicin in Patients Affected by Metastatic Small Cell Lung Carcinoma
Acronym: NGR007
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGR007; 2006-005700-14 (EudraCT Number)
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Small Cell Lung Cancer
Keywords: NGR-hTNF; SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A: NGR-hTNF + doxorubicin (Experimental): NGR-hTNF plus doxorubicin
  Interventions: Drug: NGR-hTNF; Drug: Doxorubicin

INTERVENTIONS:
Drug: NGR-hTNF — iv q3W 0.8 mcg/sqm NGR-hTNF
Drug: Doxorubicin — iv q3W 75 mg/sqm doxorubicin 60 minutes after NGR-hTNF infusion

SUMMARY:
The main objective of the trial is to document the progression free survival (PFS) in advanced or metastatic small cell lung carcinoma (SCLC) patients previously treated with at least one therapeutic regimen

DETAILED DESCRIPTION:
This is a phase II, open-label, non-randomized study that will be conducted in patients affected by advanced or metastatic SCLC, previously treated with at least one therapeutic regimen, that will be conducted using Simon's two-stage design method.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years affected by SCLC previously treated with at least one therapeutic regimen (including doxorubicin). However, in case of patient already pretreated with doxorubicin, a previous cumulative dose of doxorubicin < 300 mg/m^2 is recommended and the current treatment has to be stopped when a maximum cumulative dose of doxorubicin 550 mg/m^2 is reached.
* Cytology or histology confirmed SCLC at first diagnosis (patient with recurrent disease do not require a confirmatory biopsy to be eligible)
* Measurable disease, defined as ≥ 1 unidimensional measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by CT scan according to RECIST criteria
* ECOG Performance status 0 - 2
* Adequate baseline bone marrow, hepatic and renal function, defined as follows:

  * Neutrophils > 1.5 x 10^9/L and platelets > 100 x 10^9/L
  * Bilirubin < 1.5 x ULN
  * AST and/or ALT < 2.5 x ULN in absence of liver metastasis
  * AST and/or ALT < 5 x ULN in presence of liver metastasis
  * Serum creatinine < 1.5 x ULN
* Normal cardiac function (LVEF ≥ 55%) and absence of uncontrolled hypertension
* Patients may have had prior therapy providing the following conditions are met:

  - Chemotherapy, radiation therapy, hormonal therapy or immunotherapy: wash-out period of 28 days before start treatment

  - Surgery: wash-out period of 14 days before start treatment
* Patients must give written informed consent to participate in the study

Exclusion Criteria:

* Concurrent anticancer therapy
* Patients may not receive any other investigational agents while on study
* Patients with myocardial infarction within the last six (6) months, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Uncontrolled hypertension
* Prolonged QTc interval (congenital or acquired)
* Patient with significant peripheral vascular disease
* Previous signs of cardiotoxicity doxorubicin related
* Clinical signs of CNS involvement
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction or contraindications to human albumin preparations or to any of the excipients
* Known hypersensitivity/allergic reaction or contraindications to anthracyclines
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation. Patients - both males and females - with reproductive potential (i.e. menopausal for less than 1-year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-02-14 (Actual); Primary Completion 2010-09-22 (Actual); Study Completion 2011-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambiase, MD, Study Director — AGC Biologics S.p.A.
Locations (5):
- Italy (5):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano, Turin
  - Azienda Ospedaliera Universitaria San Martino, Genoa
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Fondazione San Raffaele del Monte Tabor, Milan

REFERENCES:
- [Derived] Gregorc V, Cavina R, Novello S, Grossi F, Lazzari C, Capelletto E, Genova C, Salini G, Lambiase A, Santoro A. NGR-hTNF and Doxorubicin as Second-Line Treatment of Patients with Small Cell Lung Cancer. Oncologist. 2018 Oct;23(10):1133-e112. doi: 10.1634/theoncologist.2018-0292. Epub 2018 Aug 3. PMID 30076277

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period: February 14th, 2007 (first enrolment), April 23rd, 2010(last enrolment); May 17th, 2011(LPLV) 5 clinical sites in Italy
Pre-assignment Details: Planned sample size n.: 27 patients; Patient screened n.:28; Patient screening failure n.: 0
Period: Overall Study
Arm/Group | A: NGR-hTNF + Doxorubicin
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: patients affected by advanced or metastatic Small Cell Lung Carcinoma (SCLC) previously treated with at least one therapeutic regimen
Groups:
- A: NGR-hTNF + Doxorubicin: NGR-hTNF plus doxorubicin
  NGR-hTNF: iv q3W 0.8 mcg/sqm
  Doxorubicin: iv q3W 75 mg/sqm doxorubicin 60 minutes after NGR-hTNF infusion
Arm/Group | A: NGR-hTNF + Doxorubicin
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62.5 [41.0 to 76.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 19
Region of Enrollment [Number; unit: participants]
  Italy | 28

OUTCOME MEASURES:

1. Primary Outcome: Antitumour Activity Defined as Progression Free Survival (PFS)
Description: Defined as the time from the date of randomization until disease progression, or death due to any cause or the last patient was known to be alive. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (Recist v1.1), as a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition the appearance of one or more new lesions was also considered progression
Time Frame: From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 150 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: NGR-hTNF + Doxorubicin
Number analyzed (Participants) | 28
months | 3.2 [1.8 to 4.7]

2. Secondary Outcome: Tumor Growth Control Rate (TGCR)
Description: evaluated according to Response evaluation criteria in solid tumors (RECIST V1.0) for target lesions and assessed by MRI:
  * Complete Response (CR):Disappearance of all target lesions
  * Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the base line sum LD
  * Progressive Disease (PD): At least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Assessed every 6-12 weeks, up to 150 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | A: NGR-hTNF + Doxorubicin
Number analyzed (Participants) | 28
Participants
  Complete Response (CR) | 0
  Partial Response(PR) | 7
  Stable disease | 8
  Progressive disease (PD) | 10
  Not assessable | 3

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time from the baseline CT scan to death due to any cause, or the last date the patient was known to be alive.
Time Frame: Through study completion, an average of 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: NGR-hTNF + Doxorubicin
Number analyzed (Participants) | 28
months | 5.6 [5.3 to 5.9]

4. Secondary Outcome: Experimental Imaging Study (DCE-MRI)
Description: To document possible modifications on vessels permeability by imaging techniques
Time Frame: during the study
Population: Though a DCE-MRI evaluation was planned by protocol for a selected number of patients, no DCE-MRI assessments were performed.
Arm/Group | A: NGR-hTNF + Doxorubicin
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Adverse Events, Reported by Severity and Relation to Treatment
Description: Evaluation according to NCI common terminology criteria for adverse events (version 3.0)
Time Frame: Through study completion, an average of 3 years
Measure: Number; unit: Event
Arm/Group | A: NGR-hTNF + Doxorubicin
Number analyzed (Participants) | 28
Event
  NGR-hTNF Related Adverse Event | 27
  Adverse Event | 349
  Serious Adverse Event | 12
  Doxorubicin AE Related Adverse Event | 206
  NGR-hTNF + Doxorubicin Related Adverse Event | 4

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 years
Arm/Group | A: NGR-hTNF + Doxorubicin
All-Cause Mortality (participants affected / at risk) | 28/28
Serious Adverse Events (participants affected / at risk) | 7/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: NGR-hTNF + Doxorubicin (N=28)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutopenia (Blood and lymphatic system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Infectious Fever (General disorders) | 1 (1)
Mucosal Inflammation (General disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: NGR-hTNF + Doxorubicin (N=28)
Aortic vlave incompetence (Cardiac disorders) | 1 (1)
Aortic valve sclerosis (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial Hypertofhy (Cardiac disorders) | 1 (1)
Bundle branch block bilateral (Cardiac disorders) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
synus tachycardia (Cardiac disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 16 (17)
Febrile neutopenia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 18 (42)
Lymphopenia (Blood and lymphatic system disorders) | 12 (15)
Neutropenia (Blood and lymphatic system disorders) | 17 (38)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (20)
Conjunctivitis (Eye disorders) | 3 (4)
Eyelid ptosis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrohea (Gastrointestinal disorders) | 4 (7)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (14)
Regurgitation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Dri Skin (Skin and subcutaneous tissue disorders) | 3 (3)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (3)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 10 (11)
Hyperurricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Metabolism acidosis (Metabolism and nutrition disorders) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Phlebitis (Vascular disorders) | 2 (2)
Asthenia (General disorders) | 5 (6)
Chills (General disorders) | 15 (20)
Extravasation (General disorders) | 1 (1)
Fatigue (General disorders) | 13 (14)
Feeling cold (General disorders) | 3 (3)
Injection site pain (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Mucosal Inflammation (General disorders) | 6 (9)
Oedema (General disorders) | 1 (1)
Pyrexia (General disorders) | 8 (8)
Wound Infection (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Respiratori tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Confusional state (Psychiatric disorders) | 2 (2)
Deprerssion (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood uric acid increased (Investigations) | 1 (2)
Blood biliribin increased (Investigations) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hipoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hypotonia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes